CLINICAL TRIAL: NCT07125807
Title: Upper Extremity Plyometric Versus Resistance Exercises to Enhance Trunk Balance in Children With Spina Bifida: A Randomized Controlled Trial
Brief Title: Plyometric vs Resistance Training for Trunk Balance in Children With Spina Bifida
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Okan University (Other)
Responsible Party: Principal Investigator, Ozgur Surenkok, Assit.Professor, Okan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 61351342/020-512
Record Dates: First submitted 2025-06-17; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Spina Bifida; Balance Changes
Keywords: Spina Bifida; Plyometric exercises; Sitting Balance; Pediatric Rehabilitation
MeSH Terms: conditions — Spinal Dysraphism

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plyometric (Experimental): plyometric exercises for trunk and sitting balance
  Interventions: Other: upper extremity plyometric exercises
- Resistance (Active Comparator): resistance exercises for trunk and sitting balance
  Interventions: Other: upper extremity resistance exercises

INTERVENTIONS:
Other: upper extremity plyometric exercises — upper extremity plyometric exercises in neuro rehabilitation
  Arms: Plyometric
Other: upper extremity resistance exercises — upper extremity resistance exercises in neuro rehabilitation
  Arms: Resistance

SUMMARY:
Objective: To compare the efficacy of upper extremity plyometric and resistance exercises in improving trunk balance in children with Spina Bifida (SB).

Methods: This randomized controlled trial (RCT) enrolled 28 children (aged 6-12 years) with lumbar-level SB, randomized to plyometric (n=14) or resistance (n=14) exercise groups for an 8-week intervention (3 days/week) alongside standard rehabilitation. Primary outcomes included Trunk Control Measurement Scale (TCMS) for static/dynamic sitting and reaching, and Pediatric Balance Scale (PBS) for overall balance. Secondary outcomes included ambulation levels via Hoffer classification.

DETAILED DESCRIPTION:
Objective:

To compare the effectiveness of upper extremity plyometric versus resistance exercises in enhancing trunk balance among children with lumbar-level Spina Bifida (SB).

Methods:

This randomized controlled trial included 28 children (aged 6-12 years) diagnosed with lumbar-level SB. Participants were randomly assigned to either a plyometric exercise group (n = 14) or a resistance exercise group (n = 14). Both groups received an 8-week intervention (three sessions per week) in addition to their standard rehabilitation programs.

Primary outcomes were assessed using the Trunk Control Measurement Scale (TCMS)-evaluating static sitting, dynamic sitting, and reaching control-and the Pediatric Balance Scale (PBS) to assess overall balance capabilities. Secondary outcomes included ambulation status, measured using the Hoffer classification.

ELIGIBILITY:
Inclusion Criteria:

* The study included children diagnosed with lumbar-level Spina Bifida,
* Aged 6 to 15 years,
* IQ of 50 or higher based on the SPARCLE cognitive assessment

Exclusion Criteria:

* History of shunt infection or revision,
* Tethered cord syndrome or syringomyelia,
* Insufficient sitting balance,
* Upper extremity spasticity or contractures,
* Severe visual or hearing impairments

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-07-20 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Trunk Control Measurement Scale (TCMS) | Day 1, right before starting treatment and right after finishing the treatment (4 weeks). using questionary scores
  It measures both static and dynamic trunk control, including selective motor control and dynamic reaching abilities. The total TCMS score ranges from 0 to 58 points. Higher scores on the TCMS indicate better trunk control and function.
Pediatric Balance Scale (PBS) | Day 1, right before starting treatment and right after finishing the treatment (4 weeks). using questionarry scores
  It is a reliable and valid clinical tool designed to assess functional balance in children aged 5 to 15 years with mild to moderate balance impairments. It is a modified version of the Berg Balance Scale tailored specifically for pediatric use, focusing on balance performance during daily functional tasks. The PBS consists of 14 items, each scored on a 5-point scale from 0 to 4: The total PBS score ranges from 0 to 56 points (14 items x 4 points each). Higher scores indicate better functional balance and motor performance.

CONTACTS AND LOCATIONS:
Locations (1):
- istanbul Okan University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No